CLINICAL TRIAL: NCT02335710
Title: In Vivo Comparison of Knee Kinematics for Subjects Implanted With a Smith & Nephew Journey Posterior Stabilizing (PS) Total Knee Arthroplasty (TKA) and Subjects Having a Normal Knee
Brief Title: Optimized Loading Response by JOURNEY II BCS Knee Increases Daily Physical Activity and Functions
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: R011373506
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Smith & Nephew Journey II BCS TKA: Subjects must be implanted with a Smith & Nephew Journey II bi-cruciate stabilizing (BCS) total knee arthroplasty (TKA) implanted by Dr. Harold Cates
  Interventions: Device: Journey II BCS TKA
- Normal knee: Subjects must have a healthy, functioning knee with no osteoarthritis or knee pathologies

INTERVENTIONS:
Device: Journey II BCS TKA
  Groups: Smith & Nephew Journey II BCS TKA

SUMMARY:
Smith & Nephew's first edition of the Journey posterior stabilizing total knee arthroplasty was analyzed by the Center for Musculoskeletal Research in a past research study, and it was determined that subjects experienced more normal-like kinematic patterns. They also achieved excessive axial rotation and a decrease in weight-bearing knee flexion. Since Smith & Nephew has made modifications to the Journey bi-cruciate stabilizing (BCS) total knee arthroplasty (TKA) design, researchers will again evaluate the kinematics of subjects implanted with the revised design to determine if subjects experience normal-like kinematic patterns and if greater weight-bearing knee flexion is achieved. The objective for this study is to analyze the in vivo kinematics for subjects implanted with a 2nd generation Journey BCS TKA and compare those patterns to subjects having a normal knee and those having the 1st generation Journey posterior stabilizing (PS) TKA that were analyzed in the previous study.

ELIGIBILITY:
Inclusion Criteria for implanted subjects:

* Implanted with a Journey II BCS
* At least 3 months post-operative with no other surgical procedures within the past 6 months
* Body Mass Index (BMI) < 40
* Body weight < 250 lbs
* Not pregnant
* Knee Society score (KSS) of > 90
* Must be able to walk on level ground without aid of any kind
* Must be able to perform deep knee bend activity without aid of any kind
* Must be able to perform chair-rise activity without aid of any kind
* Must be willing to sign both Informed Consent and HIPAA forms
* Speak English

Exclusion Criteria for implanted subjects:

* Other surgical procedures performed within the past 6 months
* < 3 months post-operative
* Pregnant
* Severe cardiopulmonary or neurologic disease
* Body weight > 250 lbs
* BMI > 40
* KSS < 90
* Unable to perform 3 required activities unassisted
* Unwilling to sign both Informed Consent and HIPAA forms
* Prisoner
* Mental disease
* Unable to speak English

Inclusion Criteria for non-implanted subjects:

* healthy, well-functioning knee with no osteoarthritis or knee pathologies
* no other surgical procedures within the past 6 months that will prohibit them from performing the three required activities
* Body Mass Index < 40
* Body weight < 250 lbs
* Not pregnant
* Knee Society score of > 90
* Must be able to walk on level ground without aid of any kind
* Must be able to perform deep knee bend activity without aid of any kind
* Must be able to perform chair-rise activity without aid of any kind
* Must be willing to sign both Informed Consent and HIPAA forms
* Speak English

Exclusion Criteria for non-implanted subjects:

* Other surgical procedures performed within the past 6 months that would prohibit them from performing three required activities
* Any past knee pathologies, osteoarthritis or knee surgeries, including implants
* Pregnant
* Severe cardiopulmonary or neurologic disease
* Body weight > 250 lbs
* BMI > 40
* KSS < 90
* Unable to perform 3 required activities unassisted
* Unwilling to sign both Informed Consent and HIPAA forms
* Prisoner
* Mental disease
* Unable to speak English

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a Smith & Nephew Journey II bi-cruciate stabilizing (BCS) implanted by Dr. Harold E. Cates or subjects with a healthy knee
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Komistek, Ph D, Principal Investigator — Employee
Locations (3):
- United States (3):
  - Tennessee Orthopaedic Clinic, Knoxville, Tennessee
  - Tennessee Orthopaedic Foundation for Education and Research, Knoxville, Tennessee
  - The University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Smith & Nephew Journey II BCS TKA: Subjects must be implanted with a Smith & Nephew Journey II BCS TKA implanted by Dr. Harold Cates
  Journey II BCS TKA
Period: Overall Study
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Started | 40 | 10
Completed | 40 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Smith & Nephew Journey II BCS TKA: Subjects must be implanted with a Smith & Nephew Journey II bi-cruciate stabilizing (BCS) total knee arthroplasty (TKA) implanted by Dr. Harold Cates
  Journey II BCS TKA
- Total: Total of all reporting groups
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee | Total
Number analyzed (Participants) | 40 | 10 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 29 | 1 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.76 (8.30) | 57.44 (7.15) | 67.29 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 6 | 33
  Male | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Kinematics Translations During Deep Knee Bend (DKB) Activity
Description: Anterior Posterior (AP) translations of medial femoral condyles during DKB Anterior Posterior (AP) translations of lateral femoral condyles during DKB
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
mm
  AP trans lateral femoral condyles 0-90 degrees | -10.11 (4.80) | -13.15 (4.78)
  AP trans medial femoral condyles 0-90 degrees | -5.15 (2.51) | -4.93 (1.78)

2. Primary Outcome: Kinematics During Deep Knee Bend (DKB) Activity
Description: Maximum weight-bearing flexion during DKB Axial Rotation (AR) during DKB
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
degrees
  Max weight-bearing flexion deep knee bend | 95.6 (20.5) | 143.6 (10.5)
  AR of the femur 0-90 degrees | 6.23 (4.44) | 17.88 (5.57)

3. Primary Outcome: Kinematics Translations During Squat to Stand (S2S) Activity
Description: Anterior Posterior (AP) translations of lateral femoral condyles during squat to stand (S2S) activity Anterior Posterior (AP) translations of medial femoral condyles during S2S
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
mm
  AP trans of lateral femoral condyle 90-0 degrees | 11.82 (4.68) | 11.30 (4.66)
  AP trans of medial femoral condyle 90-0 degrees | 5.49 (2.25) | 4.37 (2.12)

4. Primary Outcome: Kinematics During Squat to Stand (S2S) Activity
Description: Maximum weight-bearing flexion during squat to stand (S2S) activity Axial Rotation (AR) of the femur during S2S
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
degrees | -7.78 (4.92) | -15.31 (6.21)

5. Primary Outcome: Kinematics Translations During Ramp up Activity
Description: AP Translations of the Medial and Lateral Femoral Condyles During Ramp Up activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
mm
  Medial Anterior Posterior Translation 0% to 33% | 0.81 (3.05) | -1.51 (1.62)
  Medial Anterior Posterior Translation 33% to 66% | 1.21 (2.69) | 1.20 (1.15)
  Medial Anterior Posterior Translation 66% to 100% | -3.16 (3.83) | 0.63 (1.44)
  Lateral Anterior Posterior Translation 0-33% | 0.40 (1.88) | -2.72 (3.18)
  Lateral Anterior Posterior Translation 33%-66% | 1.88 (3.50) | 3.43 (2.20)
  Lateral Anterior Posterior Translation 66%-100% | -4.39 (5.63) | -2.24 (2.01)

6. Primary Outcome: Kinematics During Ramp up Activity
Description: AR of the femur during Ramp Up activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
degrees
  AR 0% to 33% | 0.50 (2.97) | 2.25 (4.15)
  AR 33% to 66% | -0.82 (2.50) | -3.64 (3.13)
  AR 66% to 100% | 1.51 (3.67) | 3.76 (3.03)

7. Primary Outcome: Kinematics Translations During Ramp Down Activity
Description: AP Translations of the Medial and Lateral Femoral Condyles during Ramp down activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
mm
  Medial Anterior Posterior Translation 0% to 33% | -0.56 (2.93) | -1.20 (1.39)
  Medial Anterior Posterior Translation 33% to 66% | -1.34 (1.94) | 0.08 (1.21)
  Medial Anterior Posterior Translation 66% to 100% | -0.35 (3.33) | 0.20 (2.25)
  Lateral Anterior Posterior Translation 0-33% | -1.45 (4.52) | -2.59 (3.56)
  Lateral Anterior Posterior Translation 33%-66% | -2.57 (3.15) | -1.85 (2.38)
  Lateral Anterior Posterior Translation 66%-100% | -0.24 (4.90) | 1.36 (2.46)

8. Primary Outcome: Kinematics During Ramp Down Activity
Description: AR of the femur during ramp down activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Number analyzed (Participants) | 40 | 10
degrees
  AR 0% to 33% | 1.10 (3.18) | 3.30 (5.15)
  AR 33% to 66% | 1.54 (3.39) | 3.04 (3.35)
  AR 66% to 100% | -0.15 (3.30) | -1.81 (3.01)

ADVERSE EVENTS:
Arm/Group | Smith & Nephew Journey II BCS TKA | Normal Knee
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/10
Other Adverse Events (participants affected / at risk) | 0/40 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes